CLINICAL TRIAL: NCT04038697
Title: Ischemic Conditioning Improves Walking Function Post Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Marquette University (Other)
Responsible Party: Principal Investigator, Matthew J. Durand, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HR-1812027206
Record Dates: First submitted 2019-07-25; First posted 2019-07-31 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Stroke, Ischemic; Stroke Hemorrhagic; Stroke, Cardiovascular
Keywords: Stroke; Rehabilitation; Ischemic Conditioning; Treadmill Training
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ischemic Conditioning + Treadmill Training (Experimental): Study participants with prior history of stroke will receive both ischemic conditioning and treadmill training.
  Interventions: Procedure: Ischemic Conditioning; Procedure: Treadmill Training
- Ischemic Conditioning Sham + Treadmill Training (Placebo Comparator): Study participants with prior history of stroke will receive both ischemic conditioning sham and treadmill training.
  Interventions: Procedure: Ischemic Conditioning Sham; Procedure: Treadmill Training
- Ischemic Conditioning Only (Active Comparator): Study participants with prior history of stroke will receive only ischemic conditioning.
  Interventions: Procedure: Ischemic Conditioning
- Healthy Control - Ischemic Conditioning + Treadmill Training (Active Comparator): Healthy control participants will receive both ischemic conditioning and treadmill training.
  Interventions: Procedure: Ischemic Conditioning; Procedure: Treadmill Training

INTERVENTIONS:
Procedure: Ischemic Conditioning — Ischemic conditioning is a well-defined, non-invasive procedure which consists of inflating a blood pressure cuff around a limb (in our study, the paretic leg), inflating the cuff to 225 mmHg to occlude blood flow to the limb for 5 minutes, releasing the cuff for 5 minutes, and repeating 5 times. In our study, participants assigned to the IC Only and IC + Treadmill Training groups will undergo twelve sessions of ischemic conditioning over a four-week period.
  Arms: Healthy Control - Ischemic Conditioning + Treadmill Training; Ischemic Conditioning + Treadmill Training; Ischemic Conditioning Only
Procedure: Ischemic Conditioning Sham — Ischemic conditioning sham consists of the same setup as ischemic conditioning, which consists of inflating a blood pressure cuff around a limb (in our study, the paretic leg), inflating the cuff to 10 mmHg for 5 minutes, releasing the cuff for 5 minutes, and repeating 5 times. 10 mmHg is a sufficient inflation pressure for study participants to perceive some cuff tightness, but is not high enough to occlude blood flow. In our study, participants assigned to the IC Sham + Treadmill Training groups will undergo twelve sessions of ischemic conditioning sham over a four-week period.
  Arms: Ischemic Conditioning Sham + Treadmill Training
Procedure: Treadmill Training — Participants will perform 3 treadmill training sessions/week for a 4 week period (12 sessions total). Treadmill training will immediately follow IC or IC Sham. Personnel performing the treadmill training will be blinded to the IC treatment group. Subjects will walk on a treadmill for six, 5-minute intervals. Walking speed will be continuously adjusted to maintain heart rate between 50% and 60% of age-adjusted heart rate reserve to minimize the confounder of intensity. If individuals cannot walk at 80% of their overground self-selected walking speed, for 5 minutes, they will be assisted into a body weight support harness. Body weight support will be adjusted (up to 50%) such that individuals can walk at 80% of their over ground walking speed for five minutes and adjusted accordingly throughout the session. Participants assigned to the Treadmill + IC and Treadmill + IC Sham groups will receive Treadmill Training.
  Arms: Healthy Control - Ischemic Conditioning + Treadmill Training; Ischemic Conditioning + Treadmill Training; Ischemic Conditioning Sham + Treadmill Training

SUMMARY:
This innovative study will address scientific and clinical areas relatively unexplored in chronic stroke that could lead to greater recovery of walking. Ischemic Conditioning (IC) is a non-invasive, simple procedure that improves motor function, exercise performance and cardiovascular function in healthy controls, but it has never been applied to the stroke population. We postulate that IC enhances the recruitment of motoneurons and results in positive neural adaptations, improves vascular endothelial function and peripheral blood flow, and together these improvements result in an increased capacity to exercise and faster walking speed. Future studies will examine the effects of IC and traditional therapy at different time points of recovery post stroke, durability of IC, molecular mechanisms of neural and cardiovascular adaptation and the efficacy compared with other adjuncts.

DETAILED DESCRIPTION:
This study will quantify the effects of Ischemic Conditioning and treadmill training on improvements in: walking speed, leg strength, neuromuscular fatigability and the hyperemic blood flow response to muscle contractions, and vascular endothelial function and aerobic exercise capacity. A randomized control design will be used with three groups of chronic stroke survivors enrolled for four weeks of training (3x/week; 12 sessions total). The groups are: IC + Treadmill Training, IC Sham + Treadmill Training, and IC only. We will also enroll a group of age- and sex-matched healthy control subjects who will undergo IC + Treadmill Training. All Aims will be tested concurrently over a five-year period. All studies will be performed in Cramer Hall at Marquette University in the Integrated Neural Engineering Rehabilitation Laboratories, the Human Performance Assessment Core, and the Physical Therapy Clinic.

Randomization of stroke patients to the three intervention groups will be performed by using randomized block designs (randomly chosen block sizes of 3, 6 and 9). This number accounts for possible dropouts and the use of non- parametric methods.

ELIGIBILITY:
Inclusion Criteria (Stroke Survivors):

1. be ≥ 1 year post diagnosis of a unilateral, cortical stroke and have residual lower extremity paresis
2. be between the ages of 18-85
3. be able to give informed consent
4. walk slower than normative values based on age and sex

Exclusion Criteria (Stroke Survivors):

1. history of deep vein thrombosis or any condition in which transient ischemia to the lower extremity is contraindicated
2. inability to follow 2 step commands
3. chronic low back or hip pain
4. history of substance abuse
5. history of head trauma
6. comorbid neurological disorder
7. any uncontrolled medical condition
8. pacemaker
9. any condition where fatiguing contractions or resisted leg contractions are contraindicated
10. inability to walk for 5 minute bouts on a treadmill with a harness supporting up to 50% of the body weight at 80% of over-ground self-selected walking speed.

Inclusion Criteria (Healthy Control Subjects):

1. be between ages of 18-85
2. be able to give informed consent

Exclusion Criteria (Healthy Control Subjects):

1. Those listed above for stroke survivors
2. History of Stroke

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Self Selected Walking Speed | Change from baseline to 4 weeks.
  We will measure how fast participants walk during the 10 meter walk test.

SECONDARY OUTCOMES:
Knee Extensor Leg Strength | Change from baseline to 4 weeks.
  Pre-treatment and after 1, 6, and 12 sessions of ischemic conditioning. We will also test 1 month post intervention
Knee Extensor Fatigability | Change from baseline to 4 weeks.
  Pre-treatment and after 1, 6, and 12 sessions of ischemic conditioning. We will also test 1 month post intervention
Flow Mediated Dilation of Non-Paretic Brachial Artery and Paretic Popliteal Artery | Change from baseline to 4 weeks.
  Pre-treatment and after 1, 6, and 12 sessions of ischemic conditioning. We will also test 1 month post intervention
Peak Oxygen Consumption | Change from baseline to 4 weeks.
  Using a recumbent bicycle and metabolic cart, we will test whole body oxygen consumption during a graded exercise test

OTHER OUTCOMES:
Six minute walk test | Change from baseline to 4 weeks.
  Clinical test for walking endurance
Lower Extremity Fugl Meyer | Change from baseline to 4 weeks.
  Clinical test for coordination
Manual Muscle Test | Change from baseline to 4 weeks.
  Clinical test for strength
Modified Ashworth Scale | Change from baseline to 4 weeks.
  Clinical test for spasticity.
  The Modified Ashworth scale measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity. Higher scores indicate worse spasticity. The scores and scale are as follows:
  0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+: Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of motion.
  2. More marked increase in muscle tone through most of the range of motion, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
Bipolar Surface Electromyography (EMG) Measurements | Change from baseline to 4 weeks.
  Bipolar surface EMG of bilateral lower extremities will be measured during walking using electrodes placed on the following muscles: rectus femoris, vastus medialis, medial hamstrings, tibialis anterior, and medial gastrocnemius.
Voluntary Activation of Paretic Muscle | Change from baseline to 4 weeks.
  Voluntary activation (neural drive to the muscle) will be assessed by stimulating the motor nerve with a brief stimulus (superimposed twitch) while the subject performs a maximal voluntary contraction (MVC).
Surface EMG Motor Unit Measurements | Change from baseline to 4 weeks.
  Surface motor unit potentials will be recorded from the vastus lateralis (VL) muscle during muscle contractions using a multi-channel linear array of 64 EMG electrodes
Hyperemic Blood Flow in Response to Muscle Contractions | Change from baseline to 4 weeks.
  Blood flow through the superficial femoral artery will be measured before and immediately after knee extensor muscle contractions using Doppler ultrasound.
Heart Rate Variability (HRV) | Change from baseline to 4 weeks.
  We will use HRV analysis to determine the effects of IC and treadmill training on sympathetic and parasympathetic control of heart rate at the same time points as above.
Step Cadence | Change from baseline to 4 weeks.
  The number of steps per minute when walking at self-selected walking speed will be measured.
Step Length | Change from baseline to 4 weeks.
  The average step length during self-selected walking speed will be measured.
Step Velocity | Change from baseline to 4 weeks.
  Step velocity, the product of cadence and step length, expressed in units of distance per time, will be measured during self-selected walking speed.
Ground Reaction Force | Change from baseline to 4 weeks.
  Ground reaction force (N) will be measured during the different phases of gait during the 10 meter walk test and reported separately.
Ankle, Hip and Knee Joint Trajectories | Change from baseline to 4 weeks.
  Ankle, hip and knee joint trajectories (Angle) will be measured separately, in both legs, during the different phases of gait during the 10 meter walk test and reported as separate values.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marquette University, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT04038697/Prot_001.pdf
  • Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT04038697/SAP_002.pdf
  • Informed Consent Form (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT04038697/ICF_000.pdf